CLINICAL TRIAL: NCT06876987
Title: The Development and Evidence Effect of a Mobile-based Situational Simulation Peritoneal Dialysis Training System in the Retraining Program of Peritoneal Dialysis Patients
Brief Title: The Mobile-based Training System in Peritoneal Dialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CMUH112-REC3-075
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Peritoneal Dialysis

STUDY DESIGN:
Intervention Model Description: The peritoneal dialysis patients participating in the study were divided into an experimental group and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine care group (Active Comparator): Receiving routine care.
  Interventions: Other: Routine care
- Retraining Program Group (Experimental): Retraining program using a mobile-based training system.
  Interventions: Other: Retraining Program

INTERVENTIONS:
Other: Routine care — Receiving routine care.
  Arms: Routine care group
Other: Retraining Program — Retraining program using a mobile-based training system.
  Arms: Retraining Program Group

SUMMARY:
The mobile-based training system can effectively improve the knowledge and technical correctness of peritoneal dialysis patients.

DETAILED DESCRIPTION:
Use mobile-based training system in peritoneal dialysis patients' retraining programs and continuously monitor the effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received peritoneal dialysis for more than 3 months; patients who have received peritoneal dialysis for less than 3 months but have recovered from peritonitis or catheter-related infection; patients who are conscious and have no mental illness.

Exclusion Criteria:

* Patients who are unable to perform peritoneal dialysis independently; illiterate; suffering from peritonitis or catheter exit site infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Peritoneal Dialysis Knowledge Scale | Immediately after recruitment, 1 month and 2 months after intervention
  Knowledge issues related to peritoneal dialysis. The Peritoneal Dialysis Care Knowledge Questionnaire will include questions related to hand hygiene, peritoneal dialysis exchange procedures, catheter exit-site care, and knowledge about infections and peritonitis. The questionnaire consists of approximately 20 questions. Each correct answer is awarded 1 point, while incorrect answers receive 0 points, with a total score of 20 points. A higher score indicates better knowledge of peritoneal dialysis care among participants.
Peritoneal Dialysis Procedure Checklist | Immediately after recruitment, 1 month and 2 months after intervention
  This scale is used to evaluate all steps involved in hand hygiene, peritoneal dialysis solution bag exchange, and catheter exit-site care. Each item is assessed with a "Yes" or "No" response, with a total of 25 items. Correct actions are awarded 1 point, while incorrect actions receive 0 points, for a maximum score of 25. Higher scores indicate better proficiency in peritoneal dialysis care-related techniques among participants.

SECONDARY OUTCOMES:
Infection event rate | 6 months after recruitment
  Infection event related to catheter exit care and peritonitis

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan